CLINICAL TRIAL: NCT01254032
Title: A 24 Week Study to Evaluate the Predictive Ability of the COPD Assessment Test (CAT) for Acute Exacerbations (PACE) in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Predictive Ability of the Chronic Obstructive Pulmonary Disease (COPD) Assessment Test (CAT) for Acute Exacerbations (PACE) in Patients With COPD
Acronym: PACE
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114169
Record Dates: First submitted 2010-12-02; First posted 2010-12-06 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: CAT; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a major health concern, with a substantial impact on a patient's life. However, the impact of COPD is currently under-recognised and, as a result, COPD is under-treated. An exacerbation of COPD is a major element that causes poor quality of life and loss of productivity. Therefore, minimizing the frequency of exacerbations is a short term treatment goal in COPD management and could improve Quality of Life (QoL) significantly in all severity groups of COPD.

Although the use of spirometry for the determination of disease severity in COPD is supported by guidelines, a lung function test alone does not provide a measurement of the overall impact of COPD on health status and is not generally available especially in primary care centre. Therefore, a standardised and effective dialogue between patients and physicians in a consultation could address the impact of COPD on a patient's QoL in this situation.

The COPD Assessment Test (CAT), recently launched in 2009, is a short and simple, self-administered questionnaire designed to assess the condition of patients and overall impact of COPD, and to improve patient-physician communication. It has been proven that the CAT has good repeatability and discriminative properties which suggest that it is sensitive to treatment effects at a group level. The CAT score with its better ability to assess the impact of COPD on patients, suggests potential to predict a significant change in COPD status such as acute exacerbations of COPD.

Since the CAT is designed to assess the impact of COPD on the patient by measuring overall impairment, it has better correlations with other instruments, such as the Clinical COPD Questionnaire (CCQ), MRC (Medical Research Council) dyspnoea scale, St George's Respiratory Questionnaire (SGRQ),and the 6-minute walk test. However, it does not correlate well with FEV1 (Forced Expiratory Volume in One Second).

While the CAT shares some similarities with other questionnaires, there are several important differences. For example, the SGRQ is substantially longer than the CAT, is complex to administer and requires the use of a computer for scoring. The CAT is designed to provide a holistic measure of the impact of COPD on the patient, whereas the MRC dyspnoea scale only measures dyspnoea, and the CCQ only assesses clinical disease control. Thus, the CAT is the only validated, short and simple assessment test which can provide a holistic measure of the impact of COPD on patients, ensuring both the physicians and the patients gain the understanding needed to manage COPD optimally.

QoL is defined as an individual's perception of their position in their life in the context of the culture and value systems. Therefore, the extent of understanding of the questionnaire might be influenced by language and ethnicities. Since the validation findings so far have been based on data from the US and Europe, PACE may provide better quality of data across ethnic groups given that mainly Asian subjects will participate in this study.

PACE is designed to evaluate whether the CAT has a high predictive value in detecting subsequent exacerbations of COPD. If so, this result might enable both patients and physicians to better target and optimise management. The primary objective is to evaluate the predictability of the CAT to have subsequent exacerbations in COPD patients. Secondary objectives are to evaluate the predictability of the CAT to have moderate to severe exacerbations or time to the first exacerbation, to identify risk predictors for COPD exacerbations, and to evaluate correlations between CAT scores and FEV1 values, or MRC dyspnea scores. An experimental objective is to evaluate the correlation between the CAT score between 2 consecutive follow-ups (e.g. Week 8 & baseline, Week 16 & Week 8) and a COPD exacerbation over the following treatment period adjusting for demographics, MRC scores, lung function parameters, medical history, and therapy history.

PACE is a multicentre, prospective, observational study designed to evaluate the predictability of the CAT score to have COPD exacerbations over 24 weeks. During the study, subjects continue taking their regular prescribed treatment. Investigators are free to make medication adjustments where required. Eligible subjects will have a clinic visit every 8 weeks, during which they will complete the CAT questionnaire, the Exacerbation Check List (ECL), MRC dyspnea scale, and spirometry. A regular phone call is placed every 8 weeks in between clinic visits to collect data for the ECL.There is no follow-up period.

550 male and female outpatient subjects will be recruited for PACE to obtain approximately 300 exacerbation events. This study will capture the winter periods in Australia, China, Korea and Taiwan, when incidence of exacerbations is at its peak.

Statistical analysis will be performed on subjects' data to derive the PACE end-points.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a major health concern, with a substantial impact on a patient's life. However, the impact of COPD is currently under-recognised and, as a result, COPD is under-treated. An exacerbation of COPD is a major element that causes poor quality of life and loss of productivity. Therefore, minimizing the frequency of exacerbations is a short term treatment goal in COPD management and could improve Quality of Life (QoL) significantly in all severity groups of COPD.

Although the use of spirometry for the determination of disease severity in COPD is supported by guidelines, a lung function test alone does not provide a measurement of the overall impact of COPD on health status and is not generally available especially in primary care centre. Therefore, a standardised and effective dialogue between patients and physicians in a consultation could address the impact of COPD on a patient's QoL in this situation.

The COPD Assessment Test (CAT), recently launched in 2009, is a short and simple, self-administered questionnaire designed to assess the condition of patients and overall impact of COPD, and to improve patient-physician communication. It has been proven that the CAT has good repeatability and discriminative properties which suggest that it is sensitive to treatment effects at a group level. The CAT score with its better ability to assess the impact of COPD on patients, suggests potential to predict a significant change in COPD status such as acute exacerbations of COPD.

Since the CAT is designed to assess the impact of COPD on the patient by measuring overall impairment, it has better correlations with other instruments, such as the Clinical COPD Questionnaire (CCQ), MRC (Medical Research Council) dyspnoea scale, St George's Respiratory Questionnaire (SGRQ),and the 6-minute walk test. However, it does not correlate well with FEV1 (Forced Expiratory Volume in One Second).

While the CAT shares some similarities with other questionnaires, there are several important differences. For example, the SGRQ is substantially longer than the CAT, is complex to administer and requires the use of a computer for scoring. The CAT is designed to provide a holistic measure of the impact of COPD on the patient, whereas the MRC dyspnoea scale only measures dyspnoea, and the CCQ only assesses clinical disease control. Thus, the CAT is the only validated, short and simple assessment test which can provide a holistic measure of the impact of COPD on patients, ensuring both the physicians and the patients gain the understanding needed to manage COPD optimally.

QoL is defined as an individual's perception of their position in their life in the context of the culture and value systems. Therefore, the extent of understanding of the questionnaire might be influenced by language and ethnicities. Since the validation findings so far have been based on data from the US and Europe, PACE may provide better quality of data across ethnic groups given that mainly Asian subjects will participate in this study.

PACE is designed to evaluate whether the CAT has a high predictive value in detecting subsequent exacerbations of COPD. If so, this result might enable both patients and physicians to better target and optimise management. The primary objective is to evaluate the predictability of the CAT to have subsequent exacerbations in COPD patients. Secondary objectives are to evaluate the predictability of the CAT to have moderate to severe exacerbations or time to the first exacerbation, to identify risk predictors for COPD exacerbations, and to evaluate correlations between CAT scores and FEV1 values, or MRC dyspnea scores. An experimental objective is to evaluate the correlation between the CAT score between 2 consecutive follow-ups (e.g. Week 8 & baseline, Week 16 & Week 8) and a COPD exacerbation over the following treatment period adjusting for demographics, MRC scores, lung function parameters, medical history, and therapy history.

PACE is a multicentre, prospective, observational study designed to evaluate the predictability of the CAT score to have COPD exacerbations over 24 weeks. During the study, subjects continue taking their regular prescribed treatment. Investigators are free to make medication adjustments where required. Eligible subjects will have a clinic visit every 8 weeks, during which they will complete the CAT questionnaire, the Exacerbation Check List (ECL), MRC dyspnea scale, and spirometry. A regular phone call is placed every 8 weeks in between clinic visits to collect data for the ECL.There is no follow-up period.

550 male and female outpatient subjects will be recruited for PACE to obtain approximately 300 exacerbation events. This study will capture the winter periods in Australia, China, Korea and Taiwan, when incidence of exacerbations is at its peak.

Statistical analysis will be performed on subjects' data to derive the PACE end-points.

For the primary endpoint, the incidence of COPD exacerbations over 24 weeks according to the baseline CAT quartiles, an adjusted model using logistic regression taking into account demographics, lung function test parameters, medical history and therapy history will be performed. This analysis also allows the risk predictors to be determined.

For quartiles of baseline CAT scores, it is expected not to have strict four equal intervals for the CAT scores since the shape of the distribution curve of the CAT scores was not linear, but sigmoidal [Jones, 2009]. The HEED data has also shown that the CAT scores were not distributed evenly. Therefore, subjects will be categorized into quartiles after the baseline CAT scores are collected to ensure an equal number of subjects in each group. The quartile 1 will be a reference group. Odds ratios will be calculated for comparing between group 1 and other groups (group 2, 3, and 4, respectively).

The above analyses will also be performed for the incidence of moderate to severe COPD exacerbations over 24 weeks and by the CAT quartiles.

Time to the first exacerbation according to the baseline CAT quartiles will be performed using Cox-regression, adjusting for demographics, lung function test parameters, medical and therapy history. Hazard ratios will be calculated for comparing between each group (group 2, 3, and 4) and group 1.

To determine the risk predictors for incidence of COPD exacerbations, a GEE (Generalised Estimating Equations, a repeated measure analysis for categorical outcomes) will be performed. A sensitivity analysis on the various dichotomized definitions for the number of COPD exacerbations (at least 1 incident, more than 1 incident, etc) will also be performed for the ROC (Receiver Operator Characteristics) and GEE analyses.

The correlation between CAT scores with FEV1 and MRC dyspnea scores will be assessed using Pearson's correlation if normality assumptions are satisfied. Otherwise the non-parametric Spearman's correlation will be presented.

ELIGIBILITY:
Inclusion Criteria:

1. Type of subject: Outpatients
2. Informed consent: Subjects must give their signed and dated written informed consent to participate.
3. Gender: Male or Female
4. Age: 40 years of age or older at Visit 1
5. COPD diagnosis: Documented diagnosis of COPD at least 6 months prior to Visit 1 in accordance with the following definition by the GOLD (Global Initiative for Chronic Obstructive Lung Disease) guideline: Post bronchodilator FEV1/FVC < 0.7.
6. History of exacerbations: At least one COPD exacerbation which required the use of any additional treatment in the last 12 months prior to Visit 1.

   For subjects who were diagnosed between 6 to 12 months prior to Visit 1, they should have at least one COPD exacerbation that required the use of any additional treatment since diagnosis.
7. Tobacco use: Smokers or ex-smokers with a smoking history of more than 10 pack years.

Exclusion Criteria:

1. Pregnancy: Women who are pregnant or lactating or are planning on becoming pregnant during the study
2. Asthma: Subjects with a current diagnosis of asthma. Subjects with a prior history of asthma are eligible if COPD is the current diagnosis.
3. Non-compliance: Subjects unable to comply with any aspect of this study protocol or scheduled visits to the study centre

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 550 male and female outpatient subjects will be enrolled in order to have approximately 300 exacerbation events. Approximately 15 centres in Korea, China, Australia, and Taiwan will be required to recruit the subjects.
  Country Planned Number of Subjects Korea 170 China 150 Taiwan 130 Australia 100
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2010-08; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Incidence of COPD exacerbations over 24 weeks according to the baseline CAT quartiles | 24 weeks

SECONDARY OUTCOMES:
Incidence of moderate to severe COPD exacerbations over 24 weeks according to the baseline CAT quartiles | 24 weeks
Time to the first exacerbation according to the baseline CAT quartiles
Risk predictors for Incidence of COPD exacerbations over 24 weeks using CAT scores, demographics, MRC scores, lung function parameters, medical history, and therapy history | 24 weeks
Correlation between the CAT scores and FEV1 values
Correlation between the CAT scores and MRC dyspnea scores

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (15):
- Australia (3):
  - GSK Investigational Site, Concord, New South Wales
  - GSK Investigational Site, Woolloongabba, Queensland
  - GSK Investigational Site, Bedford Park, South Australia
- China (7):
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Wuhan, Hubei
  - GSK Investigational Site, Suzhou, Jiangsu
  - GSK Investigational Site, Shenyang, Liaoning
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Chongqing
  - GSK Investigational Site, Shanghai
- GSK Investigational Site, Seoul, South Korea
- Taiwan (4):
  - GSK Investigational Site, Changhua
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Lee SD, Huang MS, Kang J, Lin CH, Park MJ, Oh YM, Kwon N, Jones PW, Sajkov D; Investigators of the Predictive Ability of CAT in Acute Exacerbations of COPD (PACE) Study. The COPD assessment test (CAT) assists prediction of COPD exacerbations in high-risk patients. Respir Med. 2014 Apr;108(4):600-8. doi: 10.1016/j.rmed.2013.12.014. Epub 2014 Jan 6. PMID 24456695
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 114169 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114169 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114169 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114169 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114169 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register